CLINICAL TRIAL: NCT02530008
Title: Breast Cancer 2-PREVENT Translational Center of Excellence (TCE) - Metastatic Markers of Recurrent Tumor Phenotype for Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 30113
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Women With Suspected or Confirmed Recurrent Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a cohort study of women with suspected or confirmed recurrent breast cancer, with accessible tumor by standard clinical biopsy, prior to starting a new therapy for recurrent metastatic disease. Study participants will be ascertained from the population of all persons greater than eighteen years of age receiving care at the clinical practices of the Rowan Breast Center (RBC) at the University of Pennsylvania. The overarching goal of this study is to identify the genetic and molecular markers of molecular evolution identified in patients who have progressed from a primary diagnosis of breast cancer to recurrent, metastatic disease. As an observational study, this study seeks to gather data regarding the molecular and genetic changes that a primary cancer undergoes as a patient's cancer recurs and ultimately progresses. We anticipate enrolling 600 women with recurrent breast cancer who meet eligibility requirements for this study. Participation in this study will include the following: a biopsy and blood collection, completion of the study questionnaire, an optional bone marrow aspiration, and repeat collection of blood, offer of a research biopsy and a optional bone marrow aspirate collection at each progression time point. The study participants' medical information will be updated and changes in disease status will be captured on a regular basis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed breast cancer - based upon pathology report of the primary or metastatic diagnosis
* Recurrent breast cancer (local, regional, or distant disease) - as determined by either clinical,radiological, or pathological evaluation
* Willing to undergo or provide tissue from a recent biopsy of recurrent tumor for both clinical and research testing
* Willing to undergo blood specimen collection
* Age 18 or over and are able to give informed consent

Exclusion Criteria:

* Non-metastatic breast cancer (stage I, II or III)
* Anticoagulation that cannot be interrupted for the purpose of study evaluation (patients must have normal INR and PTT at the time of study biopsy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with recurrent breast cancer
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2024-10 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
subjects with detectable DTCs/CTCs | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Angela DeMichele, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (2):
- United States (2):
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania